CLINICAL TRIAL: NCT06569368
Title: A Phase II Trial Utilizing Metronidazole to Optimize the Microbiome of Rectal Adenocarcinoma Undergoing Neoadjuvant Therapy
Brief Title: Trial Utilizing Metronidazole to Optimize the Microbiome of Rectal Adenocarcinoma Undergoing Neoadjuvant Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0880; NCI-2025-07395 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Neoadjuvant Therapy + Metronidazole (Experimental): Participants found to be eligible to take part in this study, will be randomly assigned (as in the flip of a coin) to receive standard therapy alone or standard therapy plus metronidazole.
  Participants are assigned to the metronidazole group, will also take 1 tablet of metronidazole by mouth every 8 hours for 2 weeks.
  Interventions: Drug: Metronidazole
- Standard of Care Neoadjuvant Therapy (No Intervention): Participants found to be eligible to take part in this study, will be randomly assigned (as in the flip of a coin) to receive standard therapy alone or standard therapy plus metronidazole.
  Participants in both study groups will receive their standard of care treatment, as assigned by their treating doctor outside of the research study.

INTERVENTIONS:
Drug: Metronidazole — Given by PO
  Arms: Standard of Care Neoadjuvant Therapy + Metronidazole

SUMMARY:
To learn if adding metronidazole to standard therapy can decrease populations of Fusobacterium nucleatum (F. nucleatum) and other anaerobes (small organisms that cause infections) in participants with rectal cancer receiving neoadjuvant therapy, compared to neoadjuvant therapy alone.

DETAILED DESCRIPTION:
* Primary Objectives Quantify the ability of a standard course of metronidazole to decrease populations of anaerobic bacteria from within rectal cancers in participants receiving neoadjuvant therapy.
* Secondary Objectives To observe and record augmented anti-tumor activity of metronidazole in combination with standard of care therapies. Although the clinical benefit of [this/these] drug(s) has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit, and thus the patient will be carefully monitored for tumor response in addition to safety and tolerability.

As part of the therapeutic efficacy of metronidazole in combination with standard of care therapies, overall survival and recurrence free survival will be assessed among participants enrolled in the study over the two years following study completion.

Quantify differential rates of pathologic response of tumors treated with metronidazole in combination with standard neoadjuvant therapy compared against historic controls. Those participants undergoing watch and wait protocols will not have the pathologic response and will not be included in the pathologic response assessment.

Exploratory analysis of immune and microbial infiltrates between participant matched pre and post treatment tissues (when available). This will include bacterial taxal populations along with populations of various immune cell populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants with locally advanced rectal cancers (T3, T4, or N+ disease) with decision to treat with total neoadjuvant therapy.
* No previous cycles of cytotoxic chemotherapy in management of the index tumor.
* Age ≥18 years. Because of dosing differences between pediatric and adult populations and the introduced variability with these regiments to the study's primary outcomes, participants <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%,)
* Participants must have adequate organ and marrow function as defined below:

absolute neutrophil count ≥1,000/mcL platelets ≥100,000/mcL total bilirubin ≤ institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN creatinine ≤ institutional ULN

* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with unresectable distant metastases are ineligible.
* Participants with unresectable primary tumors are ineligible.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of metronidazole on the developing human fetus are unknown. For this reason and because B2 agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Both English and non-English-speaking participants will be eligible for inclusion in the trial.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 1 year prior to entering the study.
* Participants who are receiving any other investigational agents.
* Participants with brain metastases or other unresectable metastases who would therefore not undergo standard of care proctectomy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metronidazole or other agents used in study.
* Prior history of hypersensitivity to metronidazole or other nitroimidazole derivatives.
* Concurrent treatment with disulfiram.
* Cockayne syndrome.
* Participants with uncontrolled intercurrent illness (Indicate clearly what type or extent).
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because metronidazole is a B2 agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with metronidazole, breastfeeding should be discontinued if the mother is treated with metronidazole. These potential risks may also apply to other agents used in this study.
* Participants who received cytotoxic chemotherapy within the last year are excluded from this study given known associations between chemotherapy administration and alterations in the tumoral microbiome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Michael G White, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org